CLINICAL TRIAL: NCT01219569
Title: The Effects of Sevoflurane and Propofol on Light Flashed Evoked Pupillometry
Brief Title: Effects of Sevoflurane and Propofol on Light Flashed Evoked Pupillometry
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Anesthesia, Geordie Grant, MD Associate Professor, Rutgers, The State University of New Jersey
Other Study IDs: 0120070222
Record Dates: First submitted 2009-04-01; First posted 2010-10-13 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2013-08

CONDITIONS: Blindness
Keywords: blindness; ischemic optic neuropathy
MeSH Terms: conditions — Blindness; Optic Neuropathy, Ischemic | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 2. Sevoflurane: Subjects will receive sevoflurane at 1.5% and 2.5% end tidal after steady state maintenance has been achieved and have pupillometry readings taken and every 10 minutes for 30 minute at each drug dose.
  Interventions: Drug: Sevoflurane
- 1.Propofol: 1.Subjects will receive propofol infusion and have pupillometry readings taken in both eyes after induction, after steady state maintenance has been achieved and at 30 minutes
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — Propofol infusion 120 and 160 mcg/kg/min in random sequence during the operative procedure
  Other Names: deprivan
  Groups: 1.Propofol
Drug: Sevoflurane — sevoflurane 1.5% and 2.5% end tidal in random sequence
  Other Names: Sevoflurane at 1.5 and 2.5% end tidal
  Groups: 2. Sevoflurane

SUMMARY:
This is a study to focus on the feasibility of using a monitor which may signal loss of visual function intraoperatively.

DETAILED DESCRIPTION:
The degree of a relative afferent pupillary defect (RAPD) has been correlated with the severity of an eye injury and has been shown to have prognostic significance as an indicator of retinal ischemia. Therefore light flashed evoked pupillometry (LFEP) may serve as a useful indicator of visual function. LFEP's are not known to be sensitive to anesthetics. We will measure LFEP's using different anesthetic techniques to see if there are measurable differences in the latency, amplitude and constriction velocity of the pupillary reflex. Prior to induction of anesthesia, pupillometer readings will be taken in the supine position in both eyes. The patient will be anesthetised using a standard induction technique. For maintenance of anesthesia a remifentanil infusion will be administered and supplemented by either propofol infusion (at 120 and 160 mcg/kg/min)or sevoflurane (at 1.5 and 2.5% end-tidal in random sequence. The patients will receive muscle relaxants as needed. Pupillometry readings will be taken in both eyes after induction, after steady maintenance has been achieved and every 10 minutes for 30 minutes at each drug dose.

ELIGIBILITY:
Inclusion Criteria:

* planned orthopedic surgery on the lower extremities and positioned on the back

Exclusion Criteria:

* recent bout of conjunctivitis or pink eye
* condition which inhibits the normal pupillary function of my eye

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects undergoing orthopedic surgery in the supine position
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2007-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Measure the pupil response using different anesthetic techniques | pupillometry measurements will be taken in both eyes after induction of anesthesia

SECONDARY OUTCOMES:
Measure the pupil response using different anesthetic techniques | When steady maintenance of anesthesia drug is obtained measure pupillometry response at 10 min
Measure the pupil response using different anesthetic techniques | When steady maintenance of anesthesia drug is obtaines measure pupillometry response at 20 minutes
Measure the pupil response using different anesthetic technique | When steady maintenance of anesthesia drug is obtained measure pu[illometry response at 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Geordie P. Grant, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- University Hospital, Newark, New Jersey, United States